CLINICAL TRIAL: NCT00377871
Title: Hemodynamic Performance in Stentless Heart Valves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); LivaNova (Industry); Abbott Medical Devices (Industry); Raimond and Dagmar Ringgård-Bohn's Foundation (Other); Carl og Ellen Hertz´ Legat (Unknown); Direktør Kurt Bønnelycke og hustru Grete Bønnelyckes Fond (Unknown); Jens Anker Andersen Fonden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-218/2-14
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2008-02

CONDITIONS: Heart Valve Diseases
Keywords: Stentless; Biological; aortic; heart; valve; prosthesis; artificial
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Valve design 1
  Interventions: Device: biological heart valve prosthesis
- 2 (Active Comparator): Valve design 2
  Interventions: Device: biological heart valve prosthesis
- Control (No Intervention): Healthy control

INTERVENTIONS:
Device: biological heart valve prosthesis — Two heart valve designs
  Arms: 1; 2

SUMMARY:
Hypothesis: Stentless bioprostheses will perform superior to stented bioprostheses in different hemodynamic and biomechanical parameters.

The study will investigate turbulence, flow and aortic root movement in a stentless bioprosthesis and compare it to a stented bioprosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Over 65 years old
* Submitted for aortic valve surgery
* No coronary surgery other than LIMA to LAD

Exclusion Criteria:

* Stentless valve implantation not possible
* Contraindications for MRI scan

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
turbulence | jan 2010
flow dynamics | jan 2010
aortic root dynamics | jan 2010
Effective orifice area | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Jonas A Funder, MD, Principal Investigator — Hjerte-lunge-karkirurgisk afdeling T, Skejby Sygehus
Locations (1):
- Hjerte-lunge-karkirurgisk afdeling T, Skejby Sygehus, Aarhus N, Denmark